CLINICAL TRIAL: NCT01458717
Title: Multicenter Prospective Randomized Phase II/III Study of Neoadjuvant Chemoradiation With Gemcitabine in Patients With Borderline Resectable Pancreatic Cancer
Brief Title: Neoadjuvant Chemoradiation in Patients With Borderline Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Young Jang, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BorderlinePancreas
Record Dates: First submitted 2011-10-19; First posted 2011-10-25 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreas; cancer; borderline resectable; locally advanced; resectability; chemotherapy; radiation; chemoradiation; neoadjuvant; survival; prognosis; recurrence; response rate
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Recurrence | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant (Experimental): Neoadjuvant - operation - maintenance chemotherapy
  Interventions: Drug: Neoadjuvant chemoradiation
- Upfront surgery (Active Comparator): Operation - adjuvant chemoradiation - maintenance chemotherapy
  Interventions: Procedure: Upfront surgery

INTERVENTIONS:
Drug: Neoadjuvant chemoradiation — * Neoadjuvant chemoradiation; 45Gy/25fx + 9Gy/5fx of radiation over 6 weeks with Gemcitabine 400mg/㎡
  * 4 weeks rest, re-evaluation for resectability
  * operation
  * start maintenance chemotherapy within 4~6 weeks after operation with Gemcitabine 1000mg/㎡ (D1, 8, 15) every 4 weeks, for 4 cycle
  Arms: Neoadjuvant
Procedure: Upfront surgery — * Operation at time of diagnosis
  * Adjuvant chemoradiation; 45Gy/25fx + 9Gy/5fx of radiation over 6 weeks with Gemcitabine 400mg/㎡
  * start maintenance chemotherapy within 4~6 weeks after completion of adjuvant chemoradiation with Gemcitabine 1000mg/㎡ (D1, 8, 15) every 4 weeks, for 4 cycle
  Arms: Upfront surgery

SUMMARY:
Previous reports suggest benefit of neoadjuvant chemoradiation treatment for borderline resectable pancreas cancer. This study is a multicenter prospective randomized phase II/III study of neoadjuvant chemoradiation with gemcitabine in patients with borderline resectable pancreas cancer. The study is designed in 2 arms, one with upfront surgery and the other with neoadjuvant chemoradiation therapy.

DETAILED DESCRIPTION:
Previous reports suggest benefit of neoadjuvant chemoradiation treatment for borderline resectable pancreas cancer.

This study is a multicenter prospective randomized phase II/III study of neoadjuvant chemoradiation with gemcitabine in patients with borderline resectable pancreas cancer. The study is designed in 2 arms, one with upfront surgery and the other with neoadjuvant chemoradiation therapy.

This phase 2/3 multicenter randomized controlled trial was designed to enroll 110 patients with BRPC who were randomly assigned to gemcitabine-based neoadjuvant chemoradiation treatment (54 Gray external beam radiation) followed by surgery or upfront surgery followed by chemoradiation treatment from four large-volume centers in Korea. The primary endpoint was the 2-year survival rate (2-YSR). Interim analysis was planned at the time of 50% case enrollment.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old or <75 years old
* ECOG 0-2
* biopsy proven adenocarcinoma of the pancreas
* no history of previous chemotherapy
* borderline resectable pancreas cancer
* no distant metastasis
* WBC at least 3,000/mm3 or absolute neutrophil count at least 1,500/mm3, Platelet count at least 125,000/mm3
* Bilirubin less than 2.5 mg/dL AST less than 5 times upper limit of normal
* Creatinine no greater than 1.5 times upper limit of normal
* informed consent

Exclusion Criteria:

* history of previous chemotherapy
* history of radiation at >25% area of bone marrow
* stage unspecified, with distant metastasis, recurrent pancreas cancer
* history of malignant neoplasm (except stage 0 cancer, skin in situ cancer except malignant melanoma). Patients who are NED after 5 years after treatment of malignant neoplasm can be candidate of this study
* pregnant, breast-feeding patient
* uncontrolled or active infection
* uncontrolled cardiopulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
2-year survival rate | 2-year actual survival outcome
  2-year actual survival outcome

SECONDARY OUTCOMES:
Median survival | after at least of 2-years follow up of all participants
  calculated from overall survival with Kaplan-Meier method
1-year survival rate | after at least of 1-year follow up of all participants
  1-year actual survival rate
R0 resection rate | within 3 weeks after operation
  according to pathology report after operation
curative resection rate | within 3 weeks after operation
  according to pathology report after operation
local recurrence | within at least 2-years follow up
  any point during the follow-up period
response rate after neoadjuvant chemoradiation | within 6 weeks after completion of neoadjuvant chemoradiation
  comparison of imaging study findings at pre- and post-neoadjuvant chemoradiation
efficacy of imaging study after neoadjuvant chemoradiation | within 3 weeks after operation
  comparison of pathology report and imaging study in patients who completed neoadjuvant chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Jang, M.D., Ph.D., Principal Investigator — Seoul National University College of Medicine
Locations (5):
- South Korea (5):
  - Center for Liver Cancer, National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul